CLINICAL TRIAL: NCT07250204
Title: A Study on Combined Low-pass Whole-genome and Methylome Testing of Bloody Nipple Discharge Specimens for Benign-Malignant Differentiation.
Status: Not yet recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Other Study IDs: LLHBCH2025YN-072
Record Dates: First submitted 2025-09-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Nipple Discharge
Keywords: Nipple Discharge; Bloody nipple discharge; Nipple aspirate fluid (NAF); Pathologic nipple discharge (PND); Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Galactorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — 1. Nipple aspirate fluid (NAF) and/or pathologic nipple discharge: collected by gentle suction or expressed discharge; aliquoted and stored at -80°C for cfDNA/DNA/RNA, proteomic, cytology, and biomarker analyses.
  2. Peripheral blood:
  （1）EDTA whole blood for germline DNA and buffy coat. （2）Plasma (from EDTA) for cfDNA and circulating biomarkers. （3）Serum (SST) for protein/biomarker assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant Cohort - Pathologic Nipple Discharge (DCIS/IDC): Adults (≥18 years) with unilateral, spontaneous, single-duct pathologic nipple discharge who undergo clinically indicated diagnostic surgery. Group assignment is based on postoperative breast pathology confirming malignant disease (e.g., ductal carcinoma in situ or invasive ductal carcinoma). Preoperative nipple discharge is collected for low-coverage whole-genome sequencing (fragmentomics/CNV) and genome-wide DNA methylation profiling. Usual care only; research testing does not alter management. Followed through surgery and receipt of final pathology; no protocol-mandated long-term follow-up.
- Benign Cohort - Pathologic Nipple Discharge (Papilloma/Duct Ectasia): Adults (≥18 years) with unilateral, spontaneous, single-duct pathologic nipple discharge who undergo clinically indicated diagnostic surgery. Group assignment is based on postoperative breast pathology confirming benign disease (e.g., intraductal papilloma, duct ectasia, other benign lesions). Preoperative nipple discharge is collected for low-coverage whole-genome sequencing (fragmentomics/CNV) and genome-wide DNA methylation profiling. Usual care only; research testing does not alter management. Followed through surgery and receipt of final pathology; no protocol-mandated long-term follow-up.

SUMMARY:
This is a prospective, single-center diagnostic study testing whether a new, minimally invasive analysis of nipple fluid can distinguish benign from malignant causes of pathologic nipple discharge. Many patients with bloody or blood-tinged nipple discharge undergo surgery to make a diagnosis, yet most are ultimately found to have benign disease. The investigators aim to develop a laboratory test that analyzes DNA in nipple fluid to help avoid unnecessary operations while still identifying cancers.

Approximately 30 adults with spontaneous, single-duct, unilateral bloody or serosanguinous nipple discharge who are already scheduled for standard diagnostic surgery will be enrolled at Hubei Cancer Hospital. Before surgery, the investigators will collect a small sample of nipple fluid (or gently obtain nipple aspirate fluid using a soft suction cup if needed) and one tube of blood. The investigators will analyze the fluid's DNA using two approaches: low-pass whole-genome analysis to look for copy number changes and fragmentation patterns, and genome-wide DNA methylation profiling. Surgical pathology will serve as the reference standard. Using these data, the investigators will build and validate a model to classify lesions as benign or malignant.

The primary outcome is diagnostic accuracy (area under the ROC curve, sensitivity, and specificity). Secondary outcomes include positive and negative predictive values, model calibration, subgroup performance (e.g., ductal carcinoma in situ vs invasive cancer), and an estimate of potential clinical impact (for example, how many benign cases might safely avoid surgery at a high-sensitivity threshold). Study test results will not affect current clinical care; all participants will receive usual evaluation and surgery. Risks are minimal and may include brief nipple discomfort or skin irritation from gentle suction and routine blood-draw risks (bruising, lightheadedness). There is no direct benefit to participants, but the findings may support a future noninvasive test to guide care and reduce unnecessary surgery. Data will be de-identified and stored securely. Expected enrollment is from September 2025 to May 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Spontaneous, unilateral, single-duct pathologic nipple discharge, predominantly bloody or serosanguinous, raising clinical suspicion of intraductal disease.
3. Planned diagnostic breast surgery/biopsy after specialist assessment (e.g., duct excision/microdochectomy, lumpectomy); patients who had ductoscopy but are still scheduled for surgery remain eligible.
4. Study sampling (nipple discharge and one peripheral blood tube) feasible before surgery/invasive diagnostics without delaying standard care.
5. Able and willing to provide written informed consent and allow access to surgical pathology and relevant clinical data.

Exclusion Criteria:

1. Physiologic or non-pathologic discharge (typically bilateral, multiduct, expressible only with manipulation; milky/clear/green) or galactorrhea due to endocrine/drug causes.
2. Active breast infection/inflammatory disease (e.g., abscess) as the source of discharge.
3. Prior diagnosis and treatment of breast cancer (surgery/radiation/systemic therapy).
4. Recent invasive ductal manipulation likely to confound analysis (e.g., ductoscopy, duct cannulation/irrigation), per investigator judgment.
5. Pregnant or lactating patients.
6. Significant hematologic disease/coagulopathy precluding safe sampling.
7. Inability to complete preoperative study sampling, refusal/withdrawal of consent, or poor compliance.
8. Any condition judged by investigators to compromise sample quality, data interpretation, or participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, single-center consecutive series at Hubei Cancer Hospital. Adults presenting with spontaneous, unilateral, single-duct bloody/serosanguinous nipple discharge and scheduled for diagnostic surgery/biopsy will undergo preoperative nipple-discharge collection for low-coverage whole-genome sequencing and methylome profiling. Postoperative pathology serves as the gold standard to classify benign vs malignant lesions. Enrollment is not restricted by gender identity; individuals with relevant breast anatomy who meet criteria may be included. Excludes physiologic discharge, infection, prior treated breast cancer, pregnancy/lactation, recent duct manipulation, and unsafe sampling conditions. Target sample size ≈30; no healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
AUC of the combined lcWGS-methylome model for distinguishing malignant vs benign lesions | From preoperative sampling to receipt of final surgical pathology (per participant); primary analysis at validation lock (≈0-3 months post-enrollment).
  Area under the ROC curve (AUC) with 95% CI in the independent validation cohort. Reference standard is postoperative pathology. Model integrates preoperative nipple discharge features (CNV/fragmentomics from low-coverage WGS and genome-wide DNA methylation) with a locked threshold selected on training.

SECONDARY OUTCOMES:
Sensitivity and specificity at a prespecified threshold (target sensitivity ≥95%) | Perioperative/Periprocedural: preoperative sampling (Day 0); outcome assessed at final surgical pathology report, up to 30 days postoperatively.
  Sensitivity (true positive rate) and specificity (true negative rate), with 95% confidence intervals, estimated in the independent validation cohort at a threshold fixed on the training set to target ≥95% sensitivity. Surgical pathology is the reference standard.
Positive and negative predictive values (PPV, NPV) | preoperative sampling (Day 0); outcome assessed at final surgical pathology, up to 30 days after surgery.
  PPV and NPV, with 95% confidence intervals, calculated in the independent validation cohort at the prespecified decision threshold, using surgical pathology as the reference standard.
Model calibration (calibration slope, intercept, and Hosmer-Lemeshow test) | Perioperative/Periprocedural: preoperative sampling (Day 0); outcome assessed at final surgical pathology report, up to 30 days postoperatively.
  Agreement between predicted probabilities and observed outcomes in the independent validation cohort; report calibration slope and intercept (with 95% confidence intervals) from logistic calibration, and Hosmer-Lemeshow goodness-of-fit p-value (by deciles). Reference standard: final surgical pathology.
Proportion of model-negative results in benign cases at a prespecified decision threshold (independent validation cohort) | Preoperative sampling (Day 0); outcome assessed at the time of the final surgical pathology report, up to 30 days postoperatively.
  Among participants with benign final surgical pathology, calculate the proportion with a model-negative result when applying a decision threshold prespecified on the training set to achieve >=95% sensitivity for malignancy. Report the percentage and 95% confidence interval. Reference standard: final surgical pathology.
Subgroup performance by pathology subtype and imaging status | Perioperative/Periprocedural: preoperative sampling (Day 0); outcome assessed at final surgical pathology report, up to 30 days postoperatively.
  Area under the ROC curve (AUC), sensitivity, and specificity (with 95% confidence intervals) in the independent validation cohort, stratified by pathology subtype (DCIS vs IDC) and by presence vs absence of preoperative imaging abnormalities (mammography/ultrasound/MRI). Sensitivity and specificity estimated at a prespecified threshold fixed on the training set to target ≥95% sensitivity. Reference standard: final surgical pathology.
Technical success rate and sample adequacy | Baseline (Day 0): sample collection; laboratory QC and adequacy assessed up to 14 days post-collection.
  Proportion of nipple discharge samples yielding sequencing libraries that pass prespecified QC thresholds and are analyzable; report percentage and 95% confidence interval. Summarize cfDNA yield (ng) and sequencing depth metrics (aligned reads and mean unique coverage) with medians and interquartile ranges.

OTHER OUTCOMES:
Differential genomic and methylation features associated with malignancy | Baseline (Day 0): preoperative biospecimen collection; analysis completed within 30 days post-collection; summarized at study completion (database lock), an average of 12 months.
  Number and list of significant copy-number variation (CNV) regions, fragmentomic indices, and differentially methylated regions (DMRs) that distinguish malignant vs benign, declared at FDR < 0.05; report effect sizes (e.g., log2 fold-change or odds ratios) with 95% confidence intervals. Features derived from baseline biospecimens in the training cohort. Reference standard: final surgical pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Xinhong, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD). The informed consent for this study and institutional/regulatory constraints do not permit external sharing of participant-level datasets. Aggregate results will be posted on ClinicalTrials.gov and reported in peer-reviewed publications. The study protocol, statistical analysis plan, and a CSR synopsis will be made available upon publication.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT07250204/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT07250204/ICF_001.pdf